CLINICAL TRIAL: NCT00418288
Title: The Effect of GLP-1 on Glucose Uptake in the Brain and Heart in Healthy Subjects During Hypoglycemia Assessed by Positron Emission Tomography
Brief Title: The Effect of GLP-1 on Glucose Uptake in the Brain and Heart in Healthy Men During Hypoglycemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2005-0089
Record Dates: First submitted 2007-01-03; First posted 2007-01-04 (Estimated); Last update posted 2008-06-10 (Estimated); Status verified 2008-06

CONDITIONS: Type 2 Diabetes; Stroke; Myocardial Infarction
Keywords: GLP-1; glucose metabolism; Type 2 diabetes; brain; PET
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Stroke; Myocardial Infarction | interventions — Glucagon-Like Peptide 1

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator)
  Interventions: Drug: glucagon-like-peptide-1
- P (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: glucagon-like-peptide-1 — intravenous infusion of 1.2pmol/kg/min for 7 hours
  Arms: A
Drug: placebo — intravenous infusion of 1.2pmol/kg/min
  Arms: P

SUMMARY:
Type 2 diabetes mellitus, T2D is a disease characterized by an immense growing prevalence world wide with an increased risk of myocardial infarction and stroke. GLP-1 has convincing effects on the high glucose levels in type 2 diabetic patients and is well tolerated. New animal studies indicate a protective effect of GLP-1 in the brain and the heart. The mechanism behind this is yet not known.

The study hypothesis is that during hypoglycaemia GLP-1 will stimulate glucose-uptake in the brain and heart independent of insulin and thereby exert protective effects in the brain.

DETAILED DESCRIPTION:
Type 2 diabetes mellitus, T2D is a disease characterized by an immense growing prevalence world wide. T2D is associated with a three-fold increase in cardiovascular complications (myocardial infarction and stroke) leading to significantly higher morbidity and mortality in this group of patients. The prospective British Diabetes Study (UKPDS) showed that neither diet alone nor the pharmaceutical treatment utilized (Sulphonylurea, Metformin, Insulin) were able to reduce these macrovascular complications. GLP-1 (glucagon-like-peptide-1)is an incretin with convincing effects on glycaemia in type 2 diabetic patients with little or no risk of hypoglycaemia. New research in animal models has shown a potential protective effect in the brain and heart in association with ischaemic damage. The mechanism behind this protective effect is not known. During hypoglycaemia the brain lacks glucose which is the main fuel for sufficient brain function. The brain will compensate by increasing glucose uptake across the blood brain barrier and similarly in the heart.

The effect of native GLP-1 on glucose uptake in the brain and heart will by visualized by fluoro-deoxy-glucose FDG-PET-scan during hypoglycaemia in healthy men. At the same time a pancreatic/pituitary clamp will be performed. The hypothesis is that GLP-1 directly will stimulate glucose uptake independent of the pancreatic hormones and through this mechanism exert neuro- and cardioprotective actions.

Comparisons: FDG-uptake in the brain and heart with GLP-1 infusion compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men
* Age 20-50 years
* Caucasian
* BMI 20-30 kg/m2

Exclusion Criteria:

* Diabetes in subject and 1.degree relatives
* Any disease of clinical relevance

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2007-01; Primary Completion 2007-10 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
The acute effect of GLP-1 on glucose uptake in the brain | 1 hour
The acute effect of GLP-1 on glucose uptake in the heart | 1 hour

SECONDARY OUTCOMES:
The acute effect of GLP-1 on glucose metabolic rate in the brain | 1 hour
The acute effect of GLP-1 on intracerebral glucose concentration | 1 hour
The acute effect of GLP-1 on lumped constant in the brain | 1 hour

CONTACTS AND LOCATIONS:
Overall Officials: Ole E Schmitz, MD, DSc, Principal Investigator — Department of pharmacology, Aarhus university
Locations (1):
- Department of pharmacology, Aarhus university, Aarhus, Denmark

REFERENCES:
- [Derived] Gejl M, Lerche S, Mengel A, Moller N, Bibby BM, Smidt K, Brock B, Sondergaard H, Botker HE, Gjedde A, Holst JJ, Hansen SB, Rungby J. Influence of GLP-1 on myocardial glucose metabolism in healthy men during normo- or hypoglycemia. PLoS One. 2014 Jan 6;9(1):e83758. doi: 10.1371/journal.pone.0083758. eCollection 2014. PMID 24400077